CLINICAL TRIAL: NCT04299711
Title: Mental Health and Its Correlates Among Chinese Adolescents Exposed to the Novel Coronavirus Disease 2019: A Longitudinal Study Protocol
Brief Title: Mental Health and Its Correlates Among Chinese Adolescents Exposed to the Novel Coronavirus Disease 2019
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Vivian SHI, Dr., University of Macau
Other Study IDs: SW888999
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Baseline: This study intends to recruit 3,428 Chinese adolescent students exposed to the novel coronavirus disease 2019 in the baseline survey
  Interventions: Other: Exposed to the novel coronavirus disease 2019
- 6-month follow-up: This study will track the mental health status among these recruited 3,428 participants exposed to the novel coronavirus disease 2019 in the 6 follow-up study.
  Interventions: Other: Exposed to the novel coronavirus disease 2019
- 12-month follow-up: This study will track the mental health status among these recruited 3,428 participants exposed to the novel coronavirus disease 2019 in the 12 follow-up study.
  Interventions: Other: Exposed to the novel coronavirus disease 2019
- 18-month follow-up: This study will track the mental health status among these recruited 3,428 participants exposed to the novel coronavirus disease 2019 in the 18 follow-up study.
  Interventions: Other: Exposed to the novel coronavirus disease 2019

INTERVENTIONS:
Other: Exposed to the novel coronavirus disease 2019 — Exposed to the novel coronavirus disease 2019

SUMMARY:
Background: Direct exposure to public health emergencies is associated with increased mental disorders. It is less clear about the prevalence of common mental disorders and its correlates in Chinese adolescents after experiencing public health emergencies.

Objective: This longitudinal study aims to estimate the prevalence of common mental disorders (i.e. depression, anxiety, and post-traumatic stress disorder) and its correlates in a sample of Chinese adolescents after experience a public health emergency, namely the novel coronavirus disease 2019 (COVID-19).

Method: This study intends to recruit 3,428 Chinese adolescent students from high and middle schools in the baseline survey. This study will track these recruited participants every 6 months via three-wave follow-up (i.e. 6-month, 12-month, and 18-month follow-ups). The demographics (e.g. age, gender, education, family background, and residence) and psychosocial factors (i.e. exposure to traumatic events, religious belief, social media exposure, loneliness, and perceived social support) associated with common mental disorders (i.e. depression, anxiety, and post-traumatic stress disorder) will be investigated in this sample population. Furthermore, a hardcopy self-report questionnaire will be disturbed to all participants. Additionally, the cross-sectional analyses will be first conducted to estimate the prevalence of mental disorders and their correlates in data of baseline survey. After obtaining the longitudinal data, the relative risk, incident rate ratios, latent class analysis, and structural equation model may be performed in this study. Missing data will be solved by the multiple imputations. Data analysis tools included the Stata 16.0 and Mplus 8.4.

Discussion: This longitudinal study will better help to understand the prevalence changes of mental disorders among Chinese adolescents following the COVID-19. These findings have the potential to provide empirical evidence about the burden of mental disease and key drivers of Chinese adolescents following the COVID-19, which can benefit the formation of public policy and mental health intervention programming. This study will close the gaps that a lack of epidemiological studies about the mental disorder prevalence and related risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. age range: 10-19;
2. full-time students in these targets high or middle schools;
3. nationality: China;
4. exposure context: COVID-19;
5. able to adequately understand the content of consent form and questionnaire;

(d) able to sufficiently state the purpose of the research and acknowledge the potential risks and benefits based on the questionnaire

Ages: 10 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will be conducted in Yibin City, Sichuan province, China. A total of six schools (two high schools and four middle schools) will be contacted for the data collection. According to the formula for the finite population for prevalence studies and the attrition rate of the cohort study, the total number of estimated sample size is 3,428, which will be recruited in the baseline study.
Sampling Method: Probability Sample
Enrollment: 3428 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
The prevalence and incidence changes of common mental disorders | 15 Oct 2020 - 15 Nov 2020
  The prevalence and incidence changes of common mental disorders (i.e. depression, anxiety, and PTSD) in a representative sample of Chinese adolescents

SECONDARY OUTCOMES:
Mental disorders and its' correlates | 15 Oct 2020 - 15 Nov 2020
  To identify demographics (e.g. age, gender, education, family background, and residence) the major psychosocial factors (i.e. exposure to traumatic events, religious belief, social media exposure, loneliness, and perceived social support) contributing to prevalence and incidence of mental disorders

IPD SHARING:
Plan to Share IPD: Undecided